CLINICAL TRIAL: NCT06766760
Title: A Pilot Study of Single-port Robot-assisted Surgery Using da Vinci SP Surgical System for the Surgical Treatment for Patients With Obstructive Sleep Apnea
Brief Title: Surgical Treatment for Patients With Obstructive Sleep Apnea by Using Da Vinci SP Surgical System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 113-01382A3
Record Dates: First submitted 2024-12-17; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- OSAS with SP Da Vinci (Experimental)
  Interventions: Device: Da Vinci SP Surgical System, Model SP1098

INTERVENTIONS:
Device: Da Vinci SP Surgical System, Model SP1098 — The da Vinci SP Surgical System is intended to assist in the accurate control of the da Vinci SP endoscope and instruments during minimally invasive endoscopic abdominopelvic, thoracoscopic, transoral otolaryngology, and breast surgical procedures. The system is indicated for adult use. It is intended to be used by trained physicians in an operating room environment.

SUMMARY:
This prospective, interventional, non-randomized, single arm, clinical trial will investigate feasibility and safety of trans-oral robotic surgery using da Vinci SP Surgical System in Taiwan for the surgical treatment of OSA. All the investigators are well trained and have received proof of training after completing the training program for da Vinci SP system provided by Intuitive.

DETAILED DESCRIPTION:
This study will be conducted in Chang Gung Memorial Hospital at Linkou.

Informed consent will be provided to patient who has an indication of surgical treatment for OSA. Study participants will sign an informed consent before any study procedure begins. Eligibilities will be assessed during screening period (2 weeks) with blood test and other routine assessments. Eligible patient will undergo surgical intervention using da Vinci SP Surgical System. Post-operation follow-up will be performed at 1 week, 1 month, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or more.
2. OSA with AHI ≥ 15
3. Has failed, refuses, or is unable to tolerate CPAP therapy
4. Indication of resection of tongue base with/without other invasive surgical procedure for OSA (i.e. tongue base resection only or multi-level surgery with tongue base resection)
5. ASA physical status classification 1-2 and adequate organ function
6. Patients willing and able to comply with study protocol requirements and follow-up
7. Informed consent

Exclusion Criteria:

1. BMI>35
2. Mouth opening too narrow for TORS or trismus
3. Betel nut chewing
4. Suspicious cancer diagnosis
5. Prior head-and-neck surgery (note: prior invasive therapy for OSA allowed)
6. Other medical condition or anatomical factor not suitable for TORS, including subject with congenital malformations in the larynx, throat or tongue; 1. Subject with an American Society of Anesthesiologists (ASA) score of Grade 4 or above during preoperative evaluation
7. Active infectious disease
8. Can't follow trial-required procedures
9. Severe concomitant illness that drastically shortens life expectancy or increases risk of therapeutic interventions

   * Severe heart disease (NYHA functional class III-IV)
   * Severe lung disease (GOLD Group C-D)
10. Long-term use of anti-coagulant
11. Patients with coagulopathy
12. Emergency surgery
13. Subject for whom any additional surgeries are planned for OSA within the study period, after the surgery in which the da Vinci SP System was used
14. Subject is pregnant or suspected to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | 3 months (+60 days) post-surgery
  Success of tongue base resection without conversion to alternative surgery
Apena Hypopnea Index | 3 months (+60 days) post-surgery
  Type I PSG measurements demonstrating Apena Hypopnea Index (AHI) reduction. An AHI of < 20 events/hour and a reduction in AHI of 50% or greater from baseline levels will be defined as success, when evaluated at 3 months (+60 days) post-surgery. Although it does not meet these criteria, it can be interpreted as an "improved" result when AHI is improved after surgery.

SECONDARY OUTCOMES:
Multi-level surgery | Intraoperative
  Multi-level surgery (procedure used)
Snoring Scale | 3 months (+60 days) post-surgery
  Snoring VAS
Operative time | Intraoperative
  Operative time (first skin incision to closure of wound)
Console time | 3 months (+60 days) post-surgery
  Console time
Transfusion and estimated blood loss | 3 months (+60 days) post-surgery
  Transfusion and estimated blood loss
Length of hospital stay | 3 months (+60 days) post-surgery
  Length of hospital stay
Complication rate | 30 days
  Rate, intraoperative and/or postoperative, Clavien system
Readmission rate | 30 days
  Readmission rate
Reoperation rate | 30 days
  Reoperation rate
Perioperative mortality | 30 days
  Perioperative mortality
Volume of resected tissue | 3 months (+60 days) post-surgery
  measured using the volume displacement method
Pain score | 3 months (+60 days) post-surgery
  Pain score (VAS)
Sleepiness Scale | 3 months (+60 days) post-surgery
  Epworth Sleepiness Scale (ESS) and Stanford Sleepiness Scale (SSS) at 3 months (+60 days) post-surgery compared to baseline
Pittsburgh Sleep Quality Index (PSQI) | at 1, 3, 6 months post-surgery
  Pittsburgh Sleep Quality Index (PSQI) at 1, 3, 6 months post-surgery compared to baseline.
Adverse Events | within 3 months (+60 days) post-surgery
  Assessment of all reported adverse events (AE) within 3 months, (+60 days) post-surgery. Summarizing the incidence and frequency of all reported adverse events and categorizing them using CTCAE.

OTHER OUTCOMES:
Imaging analysis | 3 months (+60 days) post-surgery
  Imaging analysis for resected tissue volume
Percentages of sleep stages | 3 months (+60 days) post-surgery
  Percentages of sleep stages (N1, N2, N3, R), at 3 months (+60 days) post-surgery compared to baseline.
Lowest oxygen saturation (LSAT) | 3 months (+60 days) post-surgery
  Lowest oxygen saturation (LSAT), at 3 months (+60 days) post-surgery compared to baseline.
Percentages of sleep time | 3 months (+60 days) post-surgery
  Percent sleep time below 90% oxygen saturation (ST90) at 3 months (+60 days) post-surgery compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Costantino A, Sampieri C, Meliante PG, De Virgilio A, Kim SH. Transoral robotic surgery in oropharyngeal squamous cell carcinoma: A comparative study between da Vinci Single-Port and da Vinci Xi systems. Oral Oncol. 2024 Jan;148:106629. doi: 10.1016/j.oraloncology.2023.106629. Epub 2023 Nov 14. PMID 37972462
- [Result] Baptista PM, Diaz Zufiaurre N, Garaycochea O, Alcalde Navarrete JM, Moffa A, Giorgi L, Casale M, O'Connor-Reina C, Plaza G. TORS as Part of Multilevel Surgery in OSA: The Importance of Careful Patient Selection and Outcomes. J Clin Med. 2022 Feb 14;11(4):990. doi: 10.3390/jcm11040990. PMID 35207264
- [Result] Lin HC, Friedman M. Transoral robotic OSA surgery. Auris Nasus Larynx. 2021 Jun;48(3):339-346. doi: 10.1016/j.anl.2020.08.025. Epub 2020 Sep 8. PMID 32917413
- [Result] Park YM, Kim DH, Kang MS, Lim JY, Choi EC, Koh YW, Kim SH. The First Human Trial of Transoral Robotic Surgery Using a Single-Port Robotic System in the Treatment of Laryngo-Pharyngeal Cancer. Ann Surg Oncol. 2019 Dec;26(13):4472-4480. doi: 10.1245/s10434-019-07802-0. Epub 2019 Sep 9. PMID 31502020
- [Result] Holsinger FC. A flexible, single-arm robotic surgical system for transoral resection of the tonsil and lateral pharyngeal wall: Next-generation robotic head and neck surgery. Laryngoscope. 2016 Apr;126(4):864-9. doi: 10.1002/lary.25724. Epub 2015 Oct 28. PMID 26509920
- [Result] Chen MM, Orosco RK, Lim GC, Holsinger FC. Improved transoral dissection of the tongue base with a next-generation robotic surgical system. Laryngoscope. 2018 Jan;128(1):78-83. doi: 10.1002/lary.26649. Epub 2017 Jul 6. PMID 28681924
- [Result] Maurice MJ, Kaouk JH. Single-Port Robot-Assisted Perineal Prostatectomy and Pelvic Lymphadenectomy: Step-by-Step Technique in a Cadaveric Model. J Endourol. 2018 May;32(S1):S93-S96. doi: 10.1089/end.2017.0707. PMID 29774808
- [Result] Chan JYK, Tsang RK, Holsinger FC, Tong MCF, Ng CWK, Chiu PWY, Ng SSM, Wong EWY. Prospective clinical trial to evaluate safety and feasibility of using a single port flexible robotic system for transoral head and neck surgery. Oral Oncol. 2019 Jul;94:101-105. doi: 10.1016/j.oraloncology.2019.05.018. Epub 2019 May 28. PMID 31178203
- [Result] Holsinger FC, Magnuson JS, Weinstein GS, Chan JYK, Starmer HM, Tsang RKY, Wong EWY, Rassekh CH, Bedi N, Hong SSY, Orosco R, O'Malley BW Jr, Moore EJ. A Next-Generation Single-Port Robotic Surgical System for Transoral Robotic Surgery: Results From Prospective Nonrandomized Clinical Trials. JAMA Otolaryngol Head Neck Surg. 2019 Nov 1;145(11):1027-1034. doi: 10.1001/jamaoto.2019.2654. PMID 31536129
- [Result] Berry RB, Brooks R, Gamaldo C, Harding SM, Lloyd RM, Quan SF, Troester MT, Vaughn BV. AASM Scoring Manual Updates for 2017 (Version 2.4). J Clin Sleep Med. 2017 May 15;13(5):665-666. doi: 10.5664/jcsm.6576. No abstract available. PMID 28416048
- [Result] Sundaram S, Bridgman SA, Lim J, Lasserson TJ. Surgery for obstructive sleep apnoea. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD001004. doi: 10.1002/14651858.CD001004.pub2. PMID 16235277
- [Result] Semelka M, Wilson J, Floyd R. Diagnosis and Treatment of Obstructive Sleep Apnea in Adults. Am Fam Physician. 2016 Sep 1;94(5):355-60. PMID 27583421
- [Result] Hao W, Wang X, Fan J, Zeng Y, Ai H, Nie S, Wei Y. Association between apnea-hypopnea index and coronary artery calcification: a systematic review and meta-analysis. Ann Med. 2021 Dec;53(1):302-317. doi: 10.1080/07853890.2021.1875137. PMID 33522282
- [Result] Reutrakul S, Mokhlesi B. Obstructive Sleep Apnea and Diabetes: A State of the Art Review. Chest. 2017 Nov;152(5):1070-1086. doi: 10.1016/j.chest.2017.05.009. Epub 2017 May 17. PMID 28527878
- [Result] Punjabi NM. The epidemiology of adult obstructive sleep apnea. Proc Am Thorac Soc. 2008 Feb 15;5(2):136-43. doi: 10.1513/pats.200709-155MG. PMID 18250205
- [Result] Lee JJ, Sundar KM. Evaluation and Management of Adults with Obstructive Sleep Apnea Syndrome. Lung. 2021 Apr;199(2):87-101. doi: 10.1007/s00408-021-00426-w. Epub 2021 Mar 13. PMID 33713177
- [Result] Heinzer R, Vat S, Marques-Vidal P, Marti-Soler H, Andries D, Tobback N, Mooser V, Preisig M, Malhotra A, Waeber G, Vollenweider P, Tafti M, Haba-Rubio J. Prevalence of sleep-disordered breathing in the general population: the HypnoLaus study. Lancet Respir Med. 2015 Apr;3(4):310-8. doi: 10.1016/S2213-2600(15)00043-0. Epub 2015 Feb 12. PMID 25682233
- [Result] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Result] Cirignotta F. Classification and definition of respiratory disorders during sleep. Minerva Med. 2004 Jun;95(3):177-85. PMID 15289747
- [Result] Sher AE, Schechtman KB, Piccirillo JF. The efficacy of surgical modifications of the upper airway in adults with obstructive sleep apnea syndrome. Sleep. 1996 Feb;19(2):156-77. doi: 10.1093/sleep/19.2.156. PMID 8855039
- [Result] Berg LM, Ankjell TKS, Sun YQ, Trovik TA, Rikardsen OG, Sjogren A, Moen K, Hellem S, Bugten V. Health-Related Quality of Life and Sleep Quality after 12 Months of Treatment in Nonsevere Obstructive Sleep Apnea: A Randomized Clinical Trial with Continuous Positive Airway Pressure and Mandibular Advancement Splints. Int J Otolaryngol. 2020 Jun 30;2020:2856460. doi: 10.1155/2020/2856460. eCollection 2020. PMID 32665778
- [Result] Sin DD, Mayers I, Man GC, Pawluk L. Long-term compliance rates to continuous positive airway pressure in obstructive sleep apnea: a population-based study. Chest. 2002 Feb;121(2):430-5. doi: 10.1378/chest.121.2.430. PMID 11834653
- [Result] Weaver TE, Grunstein RR. Adherence to continuous positive airway pressure therapy: the challenge to effective treatment. Proc Am Thorac Soc. 2008 Feb 15;5(2):173-8. doi: 10.1513/pats.200708-119MG. PMID 18250209
- [Result] Vicini C, Montevecchi F. Transoral Robotic Surgery for Obstructive Sleep Apnea: Past, Present, and Future. Sleep Med Clin. 2019 Mar;14(1):67-72. doi: 10.1016/j.jsmc.2018.10.008. Epub 2018 Nov 30. PMID 30709535
- [Result] Vicini C, Montevecchi F, Campanini A, Dallan I, Hoff PT, Spector ME, Thaler E, Ahn J, Baptista P, Remacle M, Lawson G, Benazzo M, Canzi P. Clinical outcomes and complications associated with TORS for OSAHS: a benchmark for evaluating an emerging surgical technology in a targeted application for benign disease. ORL J Otorhinolaryngol Relat Spec. 2014;76(2):63-9. doi: 10.1159/000360768. Epub 2014 Apr 23. PMID 24777053
- [Result] Lin HC, Friedman M, Chang HW, Gurpinar B. The efficacy of multilevel surgery of the upper airway in adults with obstructive sleep apnea/hypopnea syndrome. Laryngoscope. 2008 May;118(5):902-8. doi: 10.1097/MLG.0b013e31816422ea. PMID 18300704
- [Result] Lan WC, Chang WD, Tsai MH, Tsou YA. Trans-oral robotic surgery versus coblation tongue base reduction for obstructive sleep apnea syndrome. PeerJ. 2019 Oct 2;7:e7812. doi: 10.7717/peerj.7812. eCollection 2019. PMID 31592178
- [Result] Tsou YA, Hsu CC, Shih LC, Lin TC, Chiu CJ, Tien VH, Tsai MH, Chang WD. Combined Transoral Robotic Tongue Base Surgery and Palate Surgery in Obstructive Sleep Apnea Syndrome: Modified Uvulopalatopharyngoplasty versus Barbed Reposition Pharyngoplasty. J Clin Med. 2021 Jul 18;10(14):3169. doi: 10.3390/jcm10143169. PMID 34300335